CLINICAL TRIAL: NCT00595140
Title: The Effect of Acute Application of Pegvisomant Alone and in Combination With Octreotide on Endogenous GH Levels During a 6 Hour Test in Patients With Acromegaly on Constant Pegvisomant Treatment
Brief Title: Acute Application of Pegvisomant and Octreotide in Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: PD Dr. Jochen Schopohl, Medizinische Klinik - Innenstadt of the University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-Nr. 2007-005585-12; EudraCT-Nr. 2007-005585-12
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-01

CONDITIONS: Acromegaly
Keywords: Acromegaly,; growth hormone receptor antagonist,; somatostatin analogue,; combined medical treatment,; acute effect,; endogenous GH
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): patients with acromegaly on stable pegvisomant therapy
  Interventions: Drug: pegvisomant
- 2 (Active Comparator): Patients with acromegaly on stable pegvisomant therapy and additional application of octreotide 100µg
  Interventions: Drug: combination with somatostatin analogue octreotide
- 3 (Active Comparator): Patients with acromegaly on stable pegvisomant therapy and additional application of cabergoline 0.5mg orally
  Interventions: Drug: combination with dopamine agonist cabergoline

INTERVENTIONS:
Drug: pegvisomant — growth hormone receptor antagonist pegvisomant in patients´ individual dose
  Other Names: Pegvisomant:; SOMAVERT 10 mg: EU/1/02/240/001; SOMAVERT 15 mg: EU/1/02/240/002; SOMAVERT 20 mg: EU/1/02/240/003; SOMAVERT 20 mg: EU/1/02/240/004
  Arms: 1
Drug: combination with somatostatin analogue octreotide — s.c., 100µg, one time
  Other Names: Octreotide: Sandostatin 100µg: MA number 29423.01.00
  Arms: 2
Drug: combination with dopamine agonist cabergoline — oral, 0.5mg, one time
  Other Names: Cabergoline: Dostinex 0.5mg: MA number 32411.00.00
  Arms: 3

SUMMARY:
The purpose of the study is to investigate the efficacy of an acute additional application of the somatostatin analogue octreotide 100µg s.c. or the dopamine agonist cabergoline 0.5mg p.o. to the receptor antagonist pegvisomant during a 6 or 9 hour profile on reducing endogenous growth hormone in patients with acromegaly on stable pegvisomant therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with acromegaly currently on stable pegvisomant therapy
* patients with diabetes mellitus may be included. Glucose levels must be controlled regularly throughout the study
* patients must not be co-treated with any other medication for acromegaly

Exclusion Criteria:

* radiotherapy within the last 2 years
* any relevant acute disease
* history of hypersensitivity against any of the used drugs
* pregnancy or lactation
* abnormal baseline findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The decrease of endogenous growth hormone | 6 or 9 hours

SECONDARY OUTCOMES:
The course of glucose, insulin and pegvisomant during the profiles | 6 or 9 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schopohl, MD, Principal Investigator — Medizinische Klinik - Innenstadt
Locations (1):
- Medizinische Klinik - Innenstadt of the University of Munich, Munich, Germany